CLINICAL TRIAL: NCT05011539
Title: Thiol-disulfide Homeostasis in Patients With Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Alaattin Karabulut, Medical Doctor, Tepecik Training and Research Hospital
Other Study IDs: TepecikTRH-AKarabulut-001
Record Dates: First submitted 2021-08-15; First posted 2021-08-18 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ovarian cancer: The patients with ovarian cancer
- Control group

SUMMARY:
Ovarian cancer is the third most common after endometrial and cervical cancer in societies with a high standard of living; It is the second most common type of gynecological cancer after cervical cancer in societies with a low standard of living, and it is also the deadliest among gynecological cancers. Dynamic thiol-disulfide homeostasis is an antioxidant system that minimizes oxidative damage and prevents cell damage. In the presence of oxidative stress, the thiol groups combine to form the disulfide structure, and when the oxidative stress condition is over, they are separated into thiol groups again. This homeostasis is impaired in conditions that cause oxidative processes such as diabetes, cardiovascular diseases, cancers, rheumatoid arthritis, and chronic kidney failure. This can be determined by measuring the total thiol and native thiol levels. Likewise, the level of ischemia modified albumin increases in the case of oxidative stress. There are studies on this homeostasis in the literature on many types of cancer; There are studies on endometrial cancer and cervical cancer, which are gynecological cancers In this study, the usability of these tests together with other diagnostic tests in the diagnosis of ovarian cancer will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological diagnosis of ovarian cancer

Exclusion Criteria:

* Having an acute or chronic disease that will cause oxidative stress
* Using alcohol/cigarettes/drugs
* Using antioxidant agents (such as vitamins A, C, E)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Ovarian cancer patients who applied to Izmir Tepecik Training and Research Hospital
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
thiol - disulfide levels | April 2021 - January 2022
  the rate of total thiol, native thiol and total oxidant/antioxidant capacity

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Tepecik Training and Research Hospital, Izmir, Konak, Turkey (Türkiye)

REFERENCES:
- [Background] Sezgin B, Kinci MF, Pirincci F, Camuzcuoglu A, Erel O, Neselioglu S, Camuzcuoglu H. Thiol-disulfide status of patients with cervical cancer. J Obstet Gynaecol Res. 2020 Nov;46(11):2423-2429. doi: 10.1111/jog.14480. Epub 2020 Sep 9. PMID 32909381